CLINICAL TRIAL: NCT00528320
Title: Clinical Evaluation of Cardiac Resynchronization Therapy With Implantable Cardioverter-defibrillator Therapy
Brief Title: Clinical Evaluation of Cardiac Resynchronization Therapy (CRT) Using the Ovatio CRT Implantable Cardioverter-defibrillator (ICD) System
Status: Approved for marketing | Type: Expanded Access
Sponsor: ELA Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ITAC06
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Congestive Heart Failure (CHF)
Keywords: Congestive Heart Failure; Heart Failure; Cardiac Resynchronization Therapy; ICD; Implantable Cardioverter-Defibrillator; Defibrillator
MeSH Terms: conditions — Heart Failure

INTERVENTIONS:
Device: Ovatio CRT

SUMMARY:
This study provides a continued access registry for cardiac resynchronization therapy with defibrillation (CRT-D), which helps to resynchronize (coordinate) the rhythm of the heart by helping the left ventricle contract (pump blood) more uniformly, in patients with severe heart failure (New York Heart Association [NYHA] Class III or IV).

Quality of life, adverse events and device success will be analyzed and reported.

DETAILED DESCRIPTION:
ICDs have been shown to increase life expectancy substantially over various drug regimens in patients with life threatening ventricular arrhythmias. Furthermore, large scale studies of cardiac resynchronization therapy in ICD-indicated heart failure patients have demonstrated improvements in functional capacity and quality of life, without unacceptable increases in morbidity or mortality.

This study provides a continued access registry for cardiac resynchronization therapy with defibrillation (CRT-D), which helps to resynchronize (coordinate) the rhythm of the heart by helping the left ventricle contract (pump blood) more uniformly, in patients with severe heart failure (NYHA Class III or IV).

Quality of life, adverse events and device success will be analyzed and reported.

ELIGIBILITY:
Inclusion Criteria:

* Accepted indication for ICD implant
* Severe heart failure (NYHA Class III or IV) at the time of enrollment
* May have pre-existing ICD, provided subject is on stable, optimal medical regime
* Sinus rhythm with spontaneous QRS duration greater than or equal to 150 ms, or a QRS duration greater than or equal to 130 ms with an inter-ventricular mechanical delay (IVMD) greater than or equal to 40 ms
* Left-ventricular ejection fraction (LVEF) of 35% or less

Exclusion Criteria:

* Any generally accepted indication for standard cardiac pacing, or any contraindication for standard cardiac pacing
* Any contraindication for ICD therapy
* Currently implanted with a lead positioned in or through the coronary sinus
* Hypertrophic or obstructive cardiomyopathy
* Acute myocarditis
* Unstable coronary symptoms (unstable angina or myocardial infarction) within the last month
* Recent or planned cardiac revascularization or coronary angioplasty
* Correctable valvular disease that is the primary cause of heart failure
* Mechanical tricuspid valve
* Chronic atrial arrhythmia or cardioversion for atrial fibrillation within the past month, or paroxysmal atrial fibrillation requiring new pharmacologic therapy within the past month
* Systolic blood pressure consistently above 170 mmHg or consistently below 80 mmHg
* Supine resting heart rate exceeding 100 bpm
* Receiving continuous IV infusion of positive inotropic therapy or intermittent therapy (IV infusion) more than twice per week
* Heart transplant recipient
* Primary pulmonary disease of a severity that might limit the patient's ability to perform a treadmill test
* Serum creatinine above 3.0 mg/dL
* Serum hepatic functions at or above three times the upper normal limit
* Cerebrovascular event within the previous three months
* Inability to walk or other physical impediments which might prevent the patient from completing a maximum, symptom-limited treadmill test
* Age of less than 18 years
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult